CLINICAL TRIAL: NCT00705757
Title: The Effects of Latanoprost, Bimatoprost and Travoprost on Periocular Skin Pigmentation
Brief Title: The Effects of Xalatan, Travatan and Lumigan on Skin Pigmentation Near the Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Summa Health System (Other)
Responsible Party: Principal Investigator, Deepak P. Edward, PI, Summa Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pfizer GA6111AX
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-12

CONDITIONS: Glaucoma; Application Site Pigmentation Changes
Keywords: periocular skin pigmentation; Lumigan; Travatan; Xalatan; latanoprost; bimatoprost; travoprost
MeSH Terms: conditions — Glaucoma | interventions — Latanoprost; Bimatoprost; Travoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lumigan (Active Comparator): Patients assigned to Lumigan/bimatoprost one drop before bedtime (qhs) to affected eye(s)
  Interventions: Drug: bimatoprost
- Xalatan (Active Comparator): Patients assigned to Xalatan/latanoprost one drop before bedtime (qhs) to affected eye(s)
  Interventions: Drug: latanoprost
- Travatan (Active Comparator): Patients assigned to Travatan/travoprost one drop before bedtime (qhs) to affected eye(s)
  Interventions: Drug: travoprost

INTERVENTIONS:
Drug: latanoprost — Xalatan/latanoprost 0.005% ophthalmic solution one drop qhs for one year
  Other Names: Xalatan 0.005%
  Arms: Xalatan
Drug: bimatoprost — Lumigan/bimatoprost 0.03% ophthalmic solution one drop qhs for one year
  Other Names: Lumigan 0.03%
  Arms: Lumigan
Drug: travoprost — Travatan/travoprost 0.004% ophthalmic solution one drop qhs for one year
  Other Names: Travatan 0.004%
  Arms: Travatan

SUMMARY:
The purpose of this study is to study changes in skin color that may be caused by using one of the three eye medicines: Xalatan, Travatan or Lumigan.

DETAILED DESCRIPTION:
One uncommon side effect of prostaglandin eye drops is a change in color of the skin around the eyes, which is reversible. There are three different brands of the medicine which are equally effective in lowering eye pressure but their likelihood of changing skin color is unknown. Qualifying patients will be randomly assigned to use one of the three eye drops. We will take skin color measurements from several locations on the face over one year to measure pigmentation changes.

ELIGIBILITY:
Inclusion Criteria:

* patients recently diagnosed with primary open angle glaucoma or ocular hypertension
* Caucasian and African American ethnicities
* Male and Female
* Age 30 and above

Exclusion Criteria:

* A history of ocular medication use within the last 12 months
* Inflammatory/ allergic skin diseases or dermatitis
* presence of periocular hyperpigmented skin lesions
* Systemic pigmentation disorders
* Use of systemic drugs that can affect skin pigmentation
* Visitation of tanning salons, or use of self tanning products
* Pregnancy or patients planning to become pregnant in the near future

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak P Edward, MD, Principal Investigator — Summa Health System; Smajo Osmanovic, MD, Principal Investigator — Arlington eye Associates
Locations (2):
- United States (2):
  - Arlington Eye Physicians, Arlington Heights, Illinois
  - Summa Health System, Akron, Ohio

REFERENCES:
- [Background] Albert DM, Gangnon RE, Zimbric ML, Damico CM, Fisher MR, Gleiser J, Grossniklaus HE, Green WR. A study of iridectomy histopathologic features of latanoprost- and non-latanoprost-treated patients. Arch Ophthalmol. 2004 Nov;122(11):1680-5. doi: 10.1001/archopht.122.11.1680. PMID 15534130
- [Background] Herndon LW, Robert D Williams, Wand M, Asrani S. Increased periocular pigmentation with ocular hypotensive lipid use in African Americans. Am J Ophthalmol. 2003 May;135(5):713-5. doi: 10.1016/s0002-9394(02)02146-3. PMID 12719085
- [Background] Kook MS, Lee K. Increased eyelid pigmentation associated with use of latanoprost. Am J Ophthalmol. 2000 Jun;129(6):804-6. doi: 10.1016/s0002-9394(00)00402-5. PMID 10926995
- [Background] Wand M, Ritch R, Isbey EK Jr, Zimmerman TJ. Latanoprost and periocular skin color changes. Arch Ophthalmol. 2001 Apr;119(4):614-5. No abstract available. PMID 11296032
- [Background] Kapur R, Osmanovic S, Toyran S, Edward DP. Bimatoprost-induced periocular skin hyperpigmentation: histopathological study. Arch Ophthalmol. 2005 Nov;123(11):1541-6. doi: 10.1001/archopht.123.11.1541. PMID 16286616
- [Background] Doshi M, Edward DP, Osmanovic S. Clinical course of bimatoprost-induced periocular skin changes in Caucasians. Ophthalmology. 2006 Nov;113(11):1961-7. doi: 10.1016/j.ophtha.2006.05.041. Epub 2006 Aug 28. PMID 16935336
- [Background] Wistrand PJ, Stjernschantz J, Olsson K. The incidence and time-course of latanoprost-induced iridial pigmentation as a function of eye color. Surv Ophthalmol. 1997 Feb;41 Suppl 2:S129-38. doi: 10.1016/s0039-6257(97)80020-3. PMID 9154289
- [Background] Alm A, Widengard I. Latanoprost: experience of 2-year treatment in Scandinavia. Acta Ophthalmol Scand. 2000 Feb;78(1):71-6. doi: 10.1034/j.1600-0420.2000.078001071.x. PMID 10726794
- [Background] McCarey BE, Kapik BM, Kane FE; Unoprostone Monotherapy Study Group. Low incidence of iris pigmentation and eyelash changes in 2 randomized clinical trials with unoprostone isopropyl 0.15%. Ophthalmology. 2004 Aug;111(8):1480-8. doi: 10.1016/j.ophtha.2003.11.013. PMID 15288975
- [Background] Alm A, Schoenfelder J, McDermott J. A 5-year, multicenter, open-label, safety study of adjunctive latanoprost therapy for glaucoma. Arch Ophthalmol. 2004 Jul;122(7):957-65. doi: 10.1001/archopht.122.7.957. PMID 15249358
- [Background] German EJ, Hurst MA, Wood D, Gilchrist J. A novel system for the objective classification of iris colour and its correlation with response to 1% tropicamide. Ophthalmic Physiol Opt. 1998 Mar;18(2):103-10. PMID 9692029
- [Background] Takamoto T, Schwartz B, Cantor LB, Hoop JS, Steffens T. Measurement of iris color using computerized image analysis. Curr Eye Res. 2001 Jun;22(6):412-9. doi: 10.1076/ceyr.22.6.412.5490. PMID 11584340
- [Background] Melgosa M, Rivas MJ, Gomez L, Hita E. Towards a colorimetric characterization of the human iris. Ophthalmic Physiol Opt. 2000 May;20(3):252-60. PMID 10897347
- [Background] Elbaum M, Kopf AW, Rabinovitz HS, Langley RG, Kamino H, Mihm MC Jr, Sober AJ, Peck GL, Bogdan A, Gutkowicz-Krusin D, Greenebaum M, Keem S, Oliviero M, Wang S. Automatic differentiation of melanoma from melanocytic nevi with multispectral digital dermoscopy: a feasibility study. J Am Acad Dermatol. 2001 Feb;44(2):207-18. doi: 10.1067/mjd.2001.110395. PMID 11174377
- [Background] Fullerton A, Fischer T, Lahti A, Wilhelm KP, Takiwaki H, Serup J. Guidelines for measurement of skin colour and erythema. A report from the Standardization Group of the European Society of Contact Dermatitis. Contact Dermatitis. 1996 Jul;35(1):1-10. doi: 10.1111/j.1600-0536.1996.tb02258.x. PMID 8896947
- [Background] Andreassi L, Flori L. Practical applications of cutaneous colorimetry. Clin Dermatol. 1995 Jul-Aug;13(4):369-73. doi: 10.1016/0738-081x(95)00069-r. PMID 8665445
- [Background] Dornelles S, Goldim J, Cestari T. Determination of the minimal erythema dose and colorimetric measurements as indicators of skin sensitivity to UV-B radiation. Photochem Photobiol. 2004 Jun;79(6):540-4. doi: 10.1562/yg-03-08.1. PMID 15291306
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Kreis RW, Middelkoop E, van Zuijlen PP. Colour evaluation in scars: tristimulus colorimeter, narrow-band simple reflectance meter or subjective evaluation? Burns. 2004 Mar;30(2):103-7. doi: 10.1016/j.burns.2003.09.029. PMID 15019115
- [Background] Youn JI, Park JY, Jo SJ, Rim JH, Choe YB. Assessment of the usefulness of skin phototype and skin color as the parameter of cutaneous narrow band UVB sensitivity in psoriasis patients. Photodermatol Photoimmunol Photomed. 2003 Oct;19(5):261-4. doi: 10.1034/j.1600-0781.2003.00047.x. PMID 14535897
- [Background] De Felice C, Flori ML, Pellegrino M, Toti P, Stanghellini E, Molinu A, Tosi P, Bagnoli F. Predictive value of skin color for illness severity in the high-risk newborn. Pediatr Res. 2002 Jan;51(1):100-5. doi: 10.1203/00006450-200201000-00018. PMID 11756647
- [Background] Tsai TF, Bowman PH, Jee SH, Maibach HI. Effects of glycolic acid on light-induced skin pigmentation in Asian and caucasian subjects. J Am Acad Dermatol. 2000 Aug;43(2 Pt 1):238-43. doi: 10.1067/mjd.2000.104894. PMID 10906645
- [Background] Rubegni P, Cevenini G, Barbini P, Flori ML, Fimiani M, Andreassi L. Quantitative characterization and study of the relationship between constitutive-facultative skin color and phototype in Caucasians. Photochem Photobiol. 1999 Sep;70(3):303-7. PMID 10483358
- [Background] Park SB, Suh DH, Youn JI. A long-term time course of colorimetric evaluation of ultraviolet light-induced skin reactions. Clin Exp Dermatol. 1999 Jul;24(4):315-20. doi: 10.1046/j.1365-2230.1999.00488.x. PMID 10457139
- [Background] Trujillo O, Vanezis P, Cermignani M. Photometric assessment of skin colour and lightness using a tristimulus colorimeter: reliability of inter and intra-investigator observations in healthy adult volunteers. Forensic Sci Int. 1996 Jul 31;81(1):1-10. doi: 10.1016/0379-0738(96)01939-1. PMID 8784989
- [Background] Maeda M, Kachi H, Matubara K, Mori S, Kitajima Y. Pigmentation abnormalities in systemic scleroderma examined by using a colorimeter (Choromo Meter CR-200). J Dermatol Sci. 1996 Mar;11(3):228-33. doi: 10.1016/0923-1811(95)00446-7. PMID 8785175
- [Background] Wu H, Wang H, Li H, Oshuaakey J, Xiao F, Ke Y, Xu H, Xiao J, Lu D, Parra E, Shriver M, Xiong M, Barton SA, Hewett-Emmett D, Liu W, Ji L. Skin reflectance in the Han Chinese and Tibetan populations. Hum Biol. 2001 Jun;73(3):461-6. doi: 10.1353/hub.2001.0043. PMID 11459426
- [Background] Van den Kerckhove E, Staes F, Flour M, Stappaerts K, Boeckx W. Reproducibility of repeated measurements on healthy skin with Minolta Chromameter CR-300. Skin Res Technol. 2001 Feb;7(1):56-9. doi: 10.1034/j.1600-0846.2001.007001056.x. PMID 11301642
- [Background] Takiwaki H, Miyaoka Y, Skrebova N, Kohno H, Arase S. Skin reflectance-spectra and colour-value dependency on measuring-head aperture area in ordinary reflectance spectrophotometry and tristimulus colourimetry. Skin Res Technol. 2002 May;8(2):94-7. doi: 10.1034/j.1600-0846.2001.80206.x. PMID 12060473
- [Background] Lee JA, Osmanovic S, Viana MA, Kapur R, Meghpara B, Edward DP. Objective measurement of periocular pigmentation. Photodermatol Photoimmunol Photomed. 2008 Dec;24(6):285-90. doi: 10.1111/j.1600-0781.2008.00377.x. PMID 19000184

RESULTS

PARTICIPANT FLOW:
Groups:
- Lumigan: Participants were assigned to use Lumigan/bimatoprost 0.03% ophthalmic solution one drop qhs for one year in affected eye(s)
- Xalatan: Participants were assigned to use Xalatan/latanoprost 0.005% ophthalmic sol. one drop qhs for one year in affected eye(s)
- Travatan: Participants were assigned to use Travatan/travoprost 0.004% ophthalmic sol., one drop qhs for one year in affected eye(s)
Period: Overall Study
Arm/Group | Lumigan | Xalatan | Travatan
Started | 32 | 29 | 28
Completed | 19 | 21 | 17
Not Completed | 13 | 8 | 11
Not completed — Lack of Efficacy | 5 | 1 | 3
Not completed — Lost to Follow-up | 7 | 6 | 6
Not completed — Withdrawal by Subject | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumigan | Xalatan | Travatan | Total
Number analyzed (Participants) | 19 | 21 | 17 | 57
Age, Continuous [Mean (Full Range); unit: years] | 61.5 [41 to 78] | 59.2 [30 to 81] | 60.5 [39 to 73] | 60.4 [30 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 9 | 27
  Male | 9 | 13 | 8 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 4 | 10
  White | 15 | 19 | 13 | 47
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Extent of Latanoprost, Bimatoprost and Travoprost Induced Periocular Skin Hyperpigmentation Over a One Year Time Course in Newly Diagnosed Primary Open Angle and Ocular Hypertension Patients.
Description: Periocular skin color was measured with the Minolta Chroma Meter CR-400 and the L*a*b* system, also known as Commission Internationale de l'Eclairage. This is a well-accepted unit of measurement in which L* corresponds to brightness and a* and b* correspond to chromaticity.
  Measurements were taken at baseline and 1 year. Data from each time point and each location (upper and lower eyelids or cheeks/face) were averaged, and subtracted from the baseline value for that location. Six predetermined areas on and around the upper and lower eyelid and 2 areas of the face/cheek were measured.Upper and lower eyelid values were averaged and reported as single value for each location ie;-upper eyelids, lower eyelid and cheek/face. A decrease in luminance indicates increased pigmentation at the site of measurement.
Time Frame: one year
Population: Newly diagnosed glaucoma and ocular hypertension, males and females, age 30 and up, Caucasians and African Americans.
Measure: Mean (Standard Error); unit: L*a*b*
Groups:
- Xalatan: Participants were assigned to use Xalatan ophthalmic solution one drop qhs for one year in affected eye(s).
- Travatan: Participants were assigned to use Travatan ophthalmic solution one drop qhs for one year in affected eye(s).
Arm/Group | Lumigan | Xalatan | Travatan
Number analyzed (Participants) | 19 | 21 | 17
L*a*b*
  Upper Lid | -0.90 (0.67) | -1.42 (0.57) | -0.90 (0.53)
  Lower Lid | -0.37 (0.30) | 0.48 (0.40) | 0.17 (0.40)
  Cheek/Face | 0.30 (0.29) | 0.55 (0.33) | 0.51 (0.41)
Statistical Analysis 1: Comparison: Lumigan vs Xalatan vs Travatan; One way ANOVA of Upper Lid; Test type: Superiority or Other; p = 0.769, ANOVA
Statistical Analysis 2: Comparison: Lumigan vs Xalatan vs Travatan; One way ANOVA of Lower Lid; Test type: Superiority or Other; p = 0.230, ANOVA
Statistical Analysis 3: Comparison: Lumigan vs Xalatan vs Travatan; One way ANOVA of cheek/face; Test type: Superiority or Other; p = 0.851, ANOVA

ADVERSE EVENTS:
Time Frame: Data was collected for one year.
Arm/Group | Lumigan | Xalatan | Travatan
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 1/32 | 0/29 | 0/28
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lumigan (N=32) | Xalatan (N=29) | Travatan (N=28)
Recurrence of iritis at 6 week visit (Eye disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No